CLINICAL TRIAL: NCT07134842
Title: Window Studies in Glioblastoma: A Phase I Trial Investigating Neoadjuvant Ipilimumab in Newly Diagnosed Glioblastoma
Brief Title: A Study Assessing if it is Safe and Possible to Treat Brain Cancer Patients With Immunotherapy Before They Receive the Standard Treatment.
Acronym: WinGlio-ipi
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/176169
Record Dates: First submitted 2025-06-30; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma; Gliosarcoma, Adult; Glioblastoma - Category
Keywords: phase 1; immunotherapy; Brain Cancer; Glioblastoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interventional (Experimental): All patients will be treated with up to two cycles of ipilimumab prior to their standard treatment. Each cycle will last 21 days.
  Interventions: Biological: Ipilimumab (3 mg/kg)

INTERVENTIONS:
Biological: Ipilimumab (3 mg/kg) — All participants will be treated with ipilimumab (3mg/kg) for up to 2 cycles. Each cycle will last 21 days with participants receiving ipilimumab on the 1st day of the cycle.

SUMMARY:
WinGlio is a phase I study investigating neoadjuvant (before surgery) ipilimumab ( a type of immunotherapy drug) in patients with newly diagnosed glioblastoma (a form of brain cancer). Participants will receive up to 2 cycles of ipilimumab prior to the standard of care treatments for this patient group which can include debulking surgery and chemoradiation. The aim of giving the ipilimumab to the participants is to see if it is safe to treat patients with this condition with ipilimumab and also to see if the drug helps to reduce or control the patient's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Radiologically or histologically confirmed, newly diagnosed de-novo supratentorial glioblastoma (including gliosarcoma)
2. Age ≥18 years
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 (see appendix 3)
4. Clinically fit for, and appropriate to receive, neoadjuvant ipilimumab followed by standard of care treatment, based on investigator and MDT judgement
5. Adequate organ and bone marrow function:

   * Hb ≥9 g/dL
   * Neutrophils ≥1.5 x 109/L
   * Platelets ≥100 x 109/L
   * Lymphocyte count ≥1.0 x 109/L
6. Adequate renal function:

   • Creatinine clearance of ≥ 50mL/min calculated by Cockroft-Gault equation
7. Adequate liver function:

   * Bilirubin ≤ 1.5 x ULN (except for patients with known Gilbert's Syndrome who may have total bilirubin ≤ 3 x ULN)
   * Aspartate or alanine transferase (AST or ALT) ≤ 2.5 x ULN
8. Life expectancy of greater than 12 weeks
9. Willing to comply with the contraceptive requirements of the trial (see section 6.3.5)
10. Willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures
11. Written informed consent

Exclusion Criteria:

1. Known extracranial metastatic or leptomeningeal disease
2. Prior treatment for glioblastoma other than a biopsy or limited resection leaving residual disease
3. Dexamethasone dose >3mg daily (or equivalent) at the time of starting study treatment
4. Antibiotics received within 30 days prior to starting study treatment, except for prophylactic antibiotics given with surgery
5. Intratumoural or peritumoural haemorrhage deemed significant by the treating clinician
6. Active autoimmune disease apart from:

   1. Skin conditions such as psoriasis, vitiligo or alopecia not requiring systemic treatment
   2. Type 1 diabetes or thyroid disease, controlled on medication
7. Any evidence of severe or uncontrolled diseases (e.g. unstable or uncompensated respiratory, cardiac, hepatic or renal disease)
8. Known hypersensitivity to ipilimumab or any of its excipients
9. Past medical history of interstitial lung disease, idiopathic pulmonary fibrosis, drug-induced interstitial disease which required steroid treatment or any evidence of clinically active interstitial lung disease.
10. Any condition requiring systemic treatment with corticosteroids (>10mg prednisolone daily or equivalent) or other immunosuppressive medications within 14 days prior to starting study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses > 10mg daily prednisolone or equivalent are permitted in the absence of active autoimmune disease.
11. Treatment with any other investigational agent within 28 days or 5 half lives of the investigational agent (whichever is longer) prior to starting ipilimumab treatment.
12. History of previous cancer within 5 years, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and non-melanoma skin lesions
13. Positive serology for Hepatitis B defined as a positive test for HepB surface antigen (HBsAg). Note: patients who are HepB core antibody (HBcAb) positive will only be eligible for the study if the HepB virus deocyribonucleic acid (DNA) test is negative and patients are willing to undergo monthly monitoring for HBV reactivation.
14. Positive serology for Hepatitis C defined as a positive test for HCV antibody
15. Diagnosis of prior immunodeficiency or organ-transplant requiring immunosuppressive therapy or known HIV or acquired immunodeficiency syndrome (AIDS)-related illness
16. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
17. Women who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From trial registration to 3 months post ipilimumab administration
  Safety and tolerability of neoadjuvant ipilimumab as assessed by serious and non-serious adverse events, graded according to CTCAE v5.0
Overall Survival at 12 months post trial registration | From trial registration to 1 year post treatment
Feasibility of neoadjuvant ipilimumab | Upon the final patient completing treatment
  The number of patients and percentage of patients completing neoadjuvant ipilimumab regimen will be reported.
Best overall objective response rate | Through study completion, an average of 14 months

SECONDARY OUTCOMES:
Overall survival at 24 months | From date of registration up to 104 weeks
Progression Free Survival | From date of registration up to date of progression
Surgical Complications | During surgery
Treatment Compliance | Through treatment completion, an average of 42 days
  Duration on treatment will be measured from treatment start to treatment discontinuation; reasons for treatment delays, dose omissions, dose reductions and treatment discontinuation will be collected; Time to surgery will also be measured and reasons for no surgery.
Changes in Eastern Cooperative Oncology Group performance status | From baseline to end of 12 month follow up
Resection Rate | postprocedural
Patient Acceptability | Through treatment completion, average of 42 days
  Patient acceptability will be assessed as the percentage of eligible patients who decline participation in the trial, and the percentage of patients who begin the neoadjuvant ipilimumab treatment but discontinue after one cycle to opt for earlier surgery or chemotherapy.
Surgeon Acceptability | Baseline
  Surgeon acceptability will be determined by the percentage of eligible patients who are not enrolled in the trial due to a surgeon's decision.
Delay in Surgery | Date of registration to date of surgery
  Delay in surgery will be defined as the time from trial registration to the date of surgery, with a focus on identifying any delays that may result from participation in the neoadjuvant treatment arm.
Changes in Health Related Quality of Life (HRQoL) as measure by EORTC QLQ-C30 and QLQ-BN20 | Screening to 3 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Paul Mulholland, MBBS, PhD, Principal Investigator — University College, London
Locations (1):
- University College London Hospital, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No